CLINICAL TRIAL: NCT04226547
Title: Clinical Trial of Atrial Fibrillation Patients Comparing Left Atrial Appendage Occlusion Therapy to Non-vitamin K Antagonist Oral Anticoagulants
Brief Title: Amplatzer Amulet LAAO vs. NOAC
Acronym: CATALYST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10310
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device Group (Experimental): Randomized to Amplatzer Amulet LAA occluder
  Interventions: Device: Left Atrial Appendage Occlusion (Amplatzer Amulet LAA Occluder)
- Control Group (Active Comparator): Randomized to NOAC
  Interventions: Drug: Non-Vitamin K Oral Antagonists

INTERVENTIONS:
Device: Left Atrial Appendage Occlusion (Amplatzer Amulet LAA Occluder) — Implantation of an Amplatzer Amulet left atrial appendage occluder
  Other Names: Amplatzer Amulet LAA Occluder
  Arms: Device Group
Drug: Non-Vitamin K Oral Antagonists — Initiation or continuation of a NOAC drug
  Other Names: NOAC
  Arms: Control Group

SUMMARY:
The objective of this trial is to evaluate the safety and effectiveness of the Amulet LAA occluder compared to NOAC therapy in patients with non-valvular AF at increased risk for ischemic stroke and who are recommended for long-term NOAC therapy.

The clinical investigation is a prospective, randomized, multicenter active control worldwide trial. Subjects will be randomized in a 1:1 ratio between the Amulet LAA occlusion device ("Device Group") and a commercially available NOAC medication ("Control Group"). The choice of NOAC in the Control Group will be left to study physician discretion.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal, persistent, or permanent non-valvular AF (documentation must include an electrocardiogram, Holter, or event recorder)
* At high risk of stroke or systemic embolism, defined as a CHA2DS2-VASc score of ≥ 2 for men and ≥ 3 for women
* Eligible for long-term NOAC therapy
* Able to comply with the required NOAC medication regimen if randomized to the Control Group
* Able to comply with the required medication regimen post-device implant if subject is randomized to the Device Group or subject is a Roll-in
* Able to understand, and is willing to provide, written informed consent to participate in the trial, prior to any clinical investigation related procedure or assessment
* 18 years of age or older, or the age of legal consent
* Able and willing to return for required follow-up visits and assessments

Exclusion Criteria:

* Requires long-term OAC therapy for a condition other than AF
* Planned cardiac intervention or surgery, which is invasive or requires sedation or anesthesia, within 3 months following randomization, other than study-related procedures such as LAAO and cardiac imaging (if applicable)
* Known contraindication to, or allergic to, aspirin, clopidogrel, or OAC medication use
* Indicated for P2Y12 platelet inhibitor for >1 year post-randomization
* In the opinion of the investigator, is considered at high risk for general anesthesia and general anesthesia is planned for the study procedure
* Has undergone atrial septal defect (ASD) repair or has an ASD closure device present
* Has undergone patent foramen ovale (PFO) repair or has a PFO closure device implanted
* Is implanted with a mechanical valve prosthesis
* Is implanted with an inferior vena cava filter
* History of rheumatic or congenital mitral valve heart disease
* Has any of the customary contraindications for a percutaneous catheterization procedure (e.g. subject is too small to accommodate the ICE probe (if planned) or required catheters, or subject has active infection or bleeding disorder)
* Customary contraindications for TEE/TOE (e.g., presence of esophageal varices, esophageal stricture, or history of esophageal cancer)
* Experienced stroke or transient ischemic attack (TIA) within 90 days prior to randomization or implant procedure (as applicable)
* Underwent any cardiac or non-cardiac intervention or surgery within 30 days prior to randomization
* Underwent catheter ablation for AF or atrial flutter within 60 days prior to randomization
* Experienced myocardial infarction within 90 days prior to randomization
* New York Heart Association Class IV Congestive Heart Failure
* Left ventricular ejection fraction ≤ 30% (per most recent assessment)
* Symptomatic carotid disease (defined as > 50% lumen diameter narrowing on CTA, MRA, or TCD with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is < 50% lumen diameter narrowing
* Has known intracranial atherosclerosis and/or intracranial small vessel disease (defined as 6 points on the Fazekas Scale)
* Reversible cause of AF (i.e., secondary to thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
* History of idiopathic or recurrent venous thromboembolism
* LAA is obliterated or surgically ligated
* Thrombocytopenia (defined as < 50,000 platelets per microliter (<50 x 10^9 /L)or anemia (defined as hemoglobin < 10 g/dL) requiring transfusions
* Hypersensitivity to any portion of the device material or individual components of the Amulet LAA occluder device (e.g., nickel allergy)
* Actively enrolled in, or plans to enroll in, a concurrent clinical study in which the active treatment arm may confound the results of this trial
* Is pregnant or breastfeeding, or pregnancy is planned during the course of the investigation
* Active endocarditis or other infection producing bacteremia
* Transient case of AF (i.e., never previously detected, provoked/induced by surgical or catheter manipulations, etc.)
* Severe renal failure (estimated glomerular filtration rate <30 ml/min/1.73m2), but not on dialysis
* Life expectancy is less than 2 years in the opinion of the Investigator
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the Investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2650 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Composite of ischemic stroke, systemic embolism, or cardiovascular (CV) mortality | 2 years
  non-inferiority
Major bleeding or clinically relevant non-major bleeding (CRNMB) events, excluding procedure related events | 2 years
  superiority
Composite of ischemic stroke or systemic embolism | 3 years
  non-inferiority

SECONDARY OUTCOMES:
Major bleeding or CRNMB events | 2 years
  non-inferiority
Major bleeding or CRNMB events | 2 years
  superiority
Disabling or fatal strokes | 2 years
  superiority

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Mt. Sinai Medical Center
Locations (127):
- United States (79):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - UAMS Medical Center, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - Mercy Medical Group - Cardiology, Sacramento, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Florida Cardiology - Altamonte Springs, Altamonte Springs, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - AdventHealth Florida Cardiology - Lake Mary, Lake Mary, Florida
  - NCH Healthcare System, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Florida Cardiology - Oviedo, Oviedo, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital (CardioVascular Group Lawrenceville), Lawrenceville, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Overland Park Mid America Cardiology, Overland Park, Kansas
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - St. Cloud Hospital - Central MN Heart Clinic, Saint Cloud, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Bryan Heart, Lincoln, Nebraska
  - CHI Health Creighton University Medical Center-Bergan Mercy, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - South Shore University Hospital-Northwell, Bay Shore, New York
  - Buffalo General Hospital, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Staten Island University Hospital Northwell, Staten Island, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - TriHealth Bethesda North Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Baylor All Saints Medical Center at Fort Worth, Forth Worth, Texas
  - Park Plaza Hospital, Houston, Texas
  - CHI St. Luke's Health Baylor College of Medicine Med. Ctr., Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Memorial Katy Cardiology Associates, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Heart Rhythm Associates, Shenandoah, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Monongalia General Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (4):
  - Ottawa Heart Institute, Ottawa, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal
  - CHUM, Montreal
  - Vancouver General Hospital (U of BC), Vancouver
- Czechia (2):
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Nemocnice Na Homolce, Prague
- Denmark (2):
  - Skejby University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (4):
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Institute Cardio. Paris-Sud - Institut Jacques Cartier, Massy
  - Mutualiste Montsouris, Paris
  - Hopital Haut Leveque, Pessac
- Germany (9):
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin, Brandenburg
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
  - Segeberger Kliniken GmbH, Bad Segeberg
  - St. Marien-Hospital-Bonn, Bonn
  - Cardioangiologisches Centrum am Bethanien Krankenhaus, Frankfurt
  - Klinikum der Justus-Liebig-Universität, Giessen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Internistisches Klinikum München SUD, Munich
  - Helios Klinikum Siegburg, Siegburg
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - The University of Hong Kong (Queen Mary Hospital), Hong Kong
- Italy (2):
  - Fondazione Toscana Gabriele Monasterio, Massa
  - Ospedale San Raffaele, Milan
- Japan (9):
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - Chiba University, Chiba, Chiba
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo, Tokyo
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Poland (2):
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Slaskie Centrum Chorob Serca, Zabrze
- Spain (4):
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- Switzerland (2):
  - Center Inselspital Bern, Bern
  - Stadtspital Triemli, Zurich
- The Royal Sussex County Hospital, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Hylek E, Camm AJ, Halperin JL, Diener HC, Thaler D, Schmidt B, Hara H, Huisman MV, Price MJ, Lakkireddy D, Gage R, Zhao H, Jensen TP, Quintana M, Windecker S. Left atrial appendage occlusion versus NOACs in patients with atrial fibrillation: Rationale and design of the CATALYST Trial. Am Heart J. 2026 Feb 2:107367. doi: 10.1016/j.ahj.2026.107367. Online ahead of print. PMID 41638386